CLINICAL TRIAL: NCT02117154
Title: Relationship Between HbA1c, Fasting Plasma Glucose, Post-prandial Glucose and Other Measures of Glycemic Control in Malaysian Type 2 Diabetes Mellitus Patients
Brief Title: Relationship Between HbA1c, Fasting Plasma Glucose, Post-prandial Glucose and Other Measures of Glycemic Control
Status: Completed | Type: Observational
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Other Study IDs: MEC 988.5
Record Dates: First submitted 2014-04-05; First posted 2014-04-17 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Continuous Glucose Monitoring System; HbA1c; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HbA1c, 6-day Professional CGM: 6-day Continuous Glucose Monitoring System (Medtronic iPro2 Professional CGM) will be deployed on a same patient for 3 times, which is one month apart
  Interventions: Device: 6-day Continuous Glucose Monitoring System

INTERVENTIONS:
Device: 6-day Continuous Glucose Monitoring System — performed 3 times on a patient, one month apart
  Other Names: Medtronic iPro2 Professional CGM

SUMMARY:
This study aims to evaluate relative contributions of fasting plasma glucose and postprandial glucose at various HbA1c levels using 6-day CGM. Evaluation of the relationship between HbA1c, CGM, serum fructosamine and eAG, will also be looked into.

HYPOTHESES:

1. Fasting hyperglycaemia is the main contributor in Malaysian T2DM patients with poor glycaemic control (high HbA1c), postprandial hyperglycaemia plays a more important role with lower HbA1c levels.
2. There is good correlation between HbA1c, CGM, serum fructosamine and eAG in Malaysian patients.

DETAILED DESCRIPTION:
Glycated haemoglobin (HbA1c) is formed via a non-enzymatic glycation pathway by the exposure of haemoglobin to plasma glucose. The HbA1c assay is widely used to assess glycaemic control in diabetes mellitus (DM) over a 60 to 90 day period and has been shown to correlate with the development of complications in both Type 1 (T1DM) and Type 2 diabetes mellitus (T2DM).

(A) HbA1c, Fasting Plasma Glucose and Post-prandial Glucose

Several studies have looked at the relationship between fasting glucose, post-prandial glucose and HbA1c, yielding conflicting results.

In 2001, one study examined the relationships between plasma glucose and HbA1c in 371 T2DM patients who were on lifestyle modification or oral antidiabetic drugs (OADs). These patients performed self monitoring of blood glucose (SMBG) 5 to 6 times per day (fasting, pre-meal and 2 hours post-prandial). In this study HbA1c had better correlation with pre-prandial glucose rather than postprandial hyperglycaemia.

A landmark study was carried out in 2003 using one-day, 4-point, SMBG profiles in 290 T2DM patients who were on oral anti-diabetic drugs (OAD) but not on insulin. This study suggested that in patients with HbA1c < 8.5%, post-prandial hyperglycaemia was the main contributor to excessive glucose levels. Conversely, in patients with HbA1c levels ≥ 8.5%, fasting hyperglycaemia predominated. This pattern has been proposed to reflect the natural progression of T2DM, with post-prandial hyperglycaemia occurring earlier in the course of T2DM and fasting hyperglycaemia gradually predominating with progressive β-cell failure.

This concept was challenged later, where 7-point SMBG profiles at baseline and after 24 weeks were performed in 1699 patients with T2DM (on OAD or insulin therapy) with HbA1c ˃ 7%. It found that fasting hyperglycaemia was the main contributor to overall hyperglycaemia (76-80%) from the lowest to highest HbA1c levels.

Another similar study was carried out in Taiwan in 2010 (Asian descent), with several key differences. This is important as Asian T2DM patients have been shown to have a predominantly insulin secretory defect as opposed to the insulin resistance which typifies T2DM in Caucasians. Different ethnic populations have also been shown to glycate haemoglobin at different rates. HbA1c is consistently higher in African Americans compared to non-Hispanic White, no matter if normal glucose tolerance (by 0.13-0.21%), pre-diabetes (by 0.26-0.30%) or diabetes (by 0.47%). Another key difference in the taiwanese study was the use of continuous glucose monitoring (CGM) over a 3 day period in 121 T2DM patients treated with OAD, which provided a far greater number of measured glucose values compared to SMBG. It found that post-prandial hyperglycaemia contributed significantly (80%) to overall hyperglycaemia when HbA1c was < 7%. At levels of HbA1c > 7%, the study reported that both fasting and post-prandial glucose levels made equal contributions to the overall glycaemic status.

(B) HbA1c, serum fructosamine and estimated average glucose (eAG)

Although HbA1c is regarded as the gold standard in the assessment of overall glycaemic status in diabetes mellitus, there are several limitations to its use. Factors affecting erythrocyte turnover, such as haemoglobinopathies (which are more prevalent in Asians), chronic renal failure, recent blood transfusion and erythropoietin therapy may render HbA1c unsuitable for assessing glycaemic status. In such instances, other methods for assessing glycaemic control may be used.

Fructosamine is formed when plasma glucose reacts with protein. Serum fructosamine levels have been used to indicate average glucose levels over a 2 to 3 week period. The correlation between serum fructosamine and HbA1c levels has been described in Caucasians but not in an Asian population12. It was reported that there was discordance between HbA1c and fructosamine, especially in the presence of nephropathy.

SMBG and CGM are alternatives to HbA1c in assessing chronic glycaemia. The A1c-derived Average Glucose (ADAG) study looked at 700 individuals (300 T1DM, 300 T2DM and 100 healthy individuals). HbA1c, 8-point SMBG and 48-hour CGM were assessed monthly over a 4 month period. Glucose levels accrued from SMBG and CGM were used to calculate estimated average glucose levels (eAG).The ADAG study identified a linear relationship between HbA1c and eAG over the preceding 8-12 weeks for both T1DM and T2DM patients with normal erythrocyte lifespan. One of the limitations of the ADAG study was the under-representation of Asians subjects.

By performing our study, we aim to evaluate the glycaemic profiles of T2DM patients over a wide spectrum of HbA1c, by using 6 day CGM, from Asian perspectives. We also hope to establish positive correlation among HbA1c, serum fructosamine, estimated average glucose and CGM in this group of population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Diagnosed with T2DM with stable HbA1c
* On OAD, insulin or combination therapy for a minimum of 3 months
* HbA1c ≥ 6%
* Estimated Glomerular Filtration Rate (eGFR) ≥ 60 ml/min
* Normal haemoglobin level Male: 13.0 - 18.0 g/dL Female: 11.5 - 16.5 g/dL Mean corpuscular volume (MCV): 77 - 95 femtoliters (fL) Mean corpuscular hemoglobin (MCH): 27 - 32 pg Mean corpuscular hemoglobin concentration (MCHC): 32 - 36 g/dL

Exclusion Criteria:

* Newly diagnosed T2DM (<3 months)
* T1DM patients
* Not on OAD or insulin therapy
* Hospitalized patients
* Patients with other co-morbidities, eg chronic liver disease, advanced cardiac disease, malignancy, on steroid therapy
* eGFR< 60ml /min
* Patients with anaemia
* Known haemoglobinopathies, eg alpha and beta thalassemia, sickle cell disease, Hemoglobin-E thalassemia etc
* Patients with history of blood transfusion in the preceding three months
* Patients who are likely to receive or donate blood / blood products during the study period
* Patients who are on erythropoietin therapy
* Patients who are pregnant or plan for pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from Diabetes Clinic, University of Malaya Medical Center
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Area Under The Curve for Glucose excursion | Measurement on total 24hours, total postprandial period in 24 hours and 4 hours postprandial period for each meal

SECONDARY OUTCOMES:
Measurement of HbA1c, fructosamine, Glycated albumin levels | Each test is repeated 3 times on monthly basis, ie month 0,1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: ALEXANDER TONG BOON TAN, MRCP (UK), Principal Investigator — University of Malaya Medical Center
Locations (1):
- University of Malaya Medical Center, Kuala Lumpur, Kuala Lumpur, Malaysia